CLINICAL TRIAL: NCT05081011
Title: Using an AI-based Voice Assistant to Manage Insulin in Diabetes: a Randomized-Control Trial
Brief Title: Managing Insulin With a Voice AI
Acronym: MIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kevin Schulman, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58276
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Medication Adherence
Keywords: Voice Assistant; Medication Management; Insulin Management; Smart Speaker; AI; Artificial Intelligence; Autonomous Prescriptions
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Voice Assistant Device (Experimental): Subjects have their insulin titrated by a voice assistant device for 8 weeks. The Voice Assistant Device software algorithm is used to provide daily insulin dose and titration instructions.
  Interventions: Device: Voice Assistant Device
- Control (Active Comparator): Subjects have their insulin titrated via standard of care for 8 weeks. The Voice Assistant Device is limited to providing a daily reminder to take medication.
  Interventions: Device: Voice Assistant Device

INTERVENTIONS:
Device: Voice Assistant Device — Voice AI-enabled smart speaker device delivers daily custom insulin titration instructions.
  Arms: Voice Assistant Device
Device: Voice Assistant Device — Voice AI-enabled smart speaker device delivers daily generic insulin reminders.
  Arms: Control

SUMMARY:
This study randomizes participants to have their basal insulin titrated either through standard of care or by receiving prompts through interactions with an AI-enabled smart speaker device. The primary objective of this study is to investigate the feasibility of an AI-enabled smart speaker device and whether such a device facilitates insulin titration management, increases insulin adherence and decreases time to optimal insulin dose. The secondary objective of the study is to explore whether the device improves glycemic control as defined by improvements in fasting blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes
* Patients clinically indicated to be taking daily long-acting insulin
* Patients currently taking long-acting insulin but necessitating active dose adjustments

Exclusion Criteria:

* Patients who do not speak English
* Patients who do not own a smart phone
* Patients who do not have stable wireless internet connection at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Schulman, MD, MBA, Principal Investigator — Stanford University; Ashwin Nayak, MD, Principal Investigator — Stanford University; Sharif Vakili, MD, MS, MBA, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nayak A, Vakili S, Nayak K, Nikolov M, Chiu M, Sosseinheimer P, Talamantes S, Testa S, Palanisamy S, Giri V, Schulman K. Use of Voice-Based Conversational Artificial Intelligence for Basal Insulin Prescription Management Among Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2340232. doi: 10.1001/jamanetworkopen.2023.40232. PMID 38039007

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Voice Assistant Device
Started | 18 | 21
Received Intervention as Randomized | 16 | 16
Completed | 16 | 16
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: Participants who received intervention as randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Voice Assistant Device | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (13.5) | 54.1 (12.3) | 55.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 8 | 16
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time to Optimal Insulin Dose
Description: Number of days between study start date and goal fasting sugar
Time Frame: 8 weeks
Population: Participants who received intervention as randomized
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
days | 56 [29.5 to 56] | 15 [6 to 27]
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.006, Log Rank — A p-value of 0.05 would be considered statistically significant

2. Primary Outcome: Insulin Medication Adherence
Description: Percentage of adherence to taking insulin based on logs over 8 weeks
Time Frame: 8 weeks
Population: Participants who received intervention as randomized
Measure: Mean (Standard Deviation); unit: percentage of adherance
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
percentage of adherance | 50.2 (43.0) | 82.9 (20.6)
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.01, Welch 2-sample method — A p-value of 0.05 would be considered statistically significant; Mean Difference (Final Values) = 32.7, 95% CI 2-sided [8.0 to 57.4]

3. Primary Outcome: Attitudes Toward Diabetes
Description: Change in Composite Score of Attitudes Toward Diabetes (PAID-5).
  A 5-item psychometrically validated self-report questionnaire on a 5 point Likert scale (0= not problem; 4= a serious problem). The scores of each item are summed to create an overall score (Minimum value = 0; Maximum value = 20). Higher scores denote higher levels of diabetes related distress.
Time Frame: Baseline and 8 weeks
Population: Participants who received intervention as randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 6.5 (4.9) | 8.4 (3.4)
  Change at Week 8 | 1.7 (4.4) | -1.9 (4.2)
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.03, Welch 2-sample method — A p-value of 0.05 would be considered statistically significant; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-6.8 to -0.4]

4. Primary Outcome: Attitudes Toward Health Technology
Description: Change in Composite Score of Attitudes Toward Health Technology. A 2-item self-report questionnaire on a 5 point Likert scale, scored 0 to 4. The scores are summed to create an overall score (Minimum value = 0, Maximum value = 8). Higher scores indicated more favorable attitudes toward health technology.
Time Frame: Baseline and 8 weeks
Population: Participants who received intervention as randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 6.6 (1.9) | 7.1 (1.5)
  Change at Week 8 | -1.1 (2.3) | 0.3 (1.4)
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.06, Welch 2-sample method; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.03 to 2.8]

5. Primary Outcome: Attitudes Toward Medication Adherence
Description: Change in Composite Score of Attitudes Toward Medication Adherence. A 5-item self-report questionnaire on a 5-point Likert scale (0 to 4). The scores are summed to create an overall score (Minimum value = 0, Maximum value = 20). Higher scores indicate more favorable attitudes toward medication adherence.
Time Frame: Baseline and 8 weeks
Population: Participants who received intervention as randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 13.6 (3.8) | 14.0 (4.4)
  Change at Week 8 | -0.1 (2.6) | 0.8 (4.3)
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.46, Welch 2-sample method; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.6 to 3.5]

6. Secondary Outcome: Percentage of Participants Who Achieved Glycemic Control
Description: Proportion (percentage) of participants with fasting sugar within goal at end of trial.
Time Frame: 8 weeks
Population: Participants who received intervention as randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
percentage of participants | 25.0 [8.3 to 52.6] | 81.3 [53.7 to 95.0]
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Comparison of percentage (proportion) of participants achieving glycemic control; Test type: Other; p = 0.005, 2-sample test; 2-sample test for equality of proportions with Yates continuity correction; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.21 to 0.91] — Comparison of percentage (proportion) of participants achieving glycemic control

7. Secondary Outcome: Glycemic Improvement
Description: Change in 3-day average fasting sugars between first 3 days and last 3 days of study
Time Frame: Day 3 and 8 weeks (assessed at the end of each 3 day period)
Population: Participants who received intervention as randomized
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Voice Assistant Device
Number analyzed (Participants) | 16 | 16
mg/dL
  Baseline | 145.9 (41.5) | 167.5 (53.9)
  Change at Week 8 | 23.0 (54.7) | -45.9 (45.9)
Statistical Analysis 1: Comparison: Control vs Voice Assistant Device; Test type: Other; p = 0.001, Welch 2-sample method; Mean Difference (Final Values) = -68.9, 95% CI 2-sided [-107.1 to -30.1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Control | Voice Assistant Device
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT05081011/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT05081011/SAP_002.pdf